CLINICAL TRIAL: NCT03027076
Title: Microbiome Studies of Urologic Chronic Pelvic Pain Syndrome
Brief Title: Microbiome of Urologic Chronic Pelvic Pain Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Funding for project not secured
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00089692
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Prostatitis; Chronic Prostatitis; Interstitial Cystitis; Painful Bladder Syndrome; Bladder Pain Syndrome
Keywords: prostatitis; chronic prostatitis; chronic pelvic pain syndrome; interstitial cystitis; painful bladder syndrome; bladder pain syndrome; biomarkers; biological markers; bacteria; microbiome; inflammation
MeSH Terms: conditions — Prostatitis; Cystitis, Interstitial; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — 1. Urine from male and female participants
  2. Expressed prostatic secretions (EPS) from male participants
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Men with UCPPS: Genitourinary Specimen Collection for microbiome evaluation
  Interventions: Procedure: Genitourinary Specimen Collection
- Asymptomatic Men: Genitourinary Specimen Collection for microbiome evaluation
  Interventions: Procedure: Genitourinary Specimen Collection
- Women with UCPPS: Collect midstream urine samples
  Interventions: Procedure: Collect midstream urine samples
- Asymptomatic Women: Collect midstream urine samples
  Interventions: Procedure: Collect midstream urine samples

INTERVENTIONS:
Procedure: Genitourinary Specimen Collection — Collect urethral swab, urine before prostatic massage (pre-M), urine after prostatic massage (post-M) and Expressed Prostatic Secretion (EPS)
  Groups: Asymptomatic Men; Men with UCPPS
Procedure: Collect midstream urine samples — Collect midstream urine samples
  Groups: Asymptomatic Women; Women with UCPPS

SUMMARY:
This research is being done to learn more about the bacteria that live in the genito-urinary tract in subjects with urologic chronic pelvic pain syndrome (UCPPS).

DETAILED DESCRIPTION:
This research is being done to learn more about the bacteria that live in the genito-urinary tract in subjects with urologic chronic pelvic pain syndrome (UCPPS).

A microbiome is defined as "the ecological community of commensal, symbiotic, and pathogenic microorganisms that literally share our body space." (Lederberg, 2001) The present study is designed to establish the prostate, urinary bladder and urethral microbiome in men with chronic prostatitis/chronic pelvic pain syndrome or the urinary bladder and urethral microbiome in women with interstitial cystitis/painful bladder syndrome.

The human urethra, bladder and prostate normally harbor microbial communities. The recent advent of large-scale "omics" technologies allows a detailed analysis of those communities. While current knowledge of the normal inhabitants of the human urogenital tract remains incomplete, more than 90% of patients with UCPPS report the onset of symptoms following a "urinary tract infection". The causative agents in most of those cases remain unknown, partly due to the limitations of older detection technologies that require the detection and isolation of a single microorganism for implicating it as a causative agent. Furthermore, many microbial species remain unculturable and therefore, are often undetectable using standard technology.

The current project will utilize state-of-the-art "omic" technology to detect and identify microbial species in the urethra and bladder of both men and women and the prostate of men. Additionally, the inflammatory response that accompanies those microbial communities will be characterized. Finally, the presence and number of microbial species will be correlated with the intensity of the inflammatory response and the severity of symptoms that patients with UCPPS experience.

ELIGIBILITY:
Inclusion Criteria:

* Consent: Participant has signed and dated the Informed Consent document, approved by the Johns Hopkins Medical Institutions Institutional Review Board;
* Agreement: Participant agrees to participate in study procedures;
* Age: Participant is at least 18 years of age;
* Symptom Severity: Participant reports a response of at least 8 on the Pain Domain of the NIH-Chronic Prostatitis Symptom Index (CPSI) Questionnaire;
* Duration of Symptoms: Symptoms have been present for at least 3 months within the preceding 6 months.

Exclusion Criteria:

* Urethral conditions: Participant has an ongoing symptomatic urethral stricture;
* Bladder conditions: Participant has a history of cystitis caused by tuberculosis, radiation therapy or cytoxan/cyclophosphamide therapy, augmentation cystoplasty or cystectomy;
* Testicular conditions: Participant diagnosed with unilateral orchialgia, without pelvic symptoms;
* Prostate conditions or procedures: Participant has a history of transurethral microwave thermotherapy (TUMT), transurethral needle ablation (TUNA), balloon dilation, prostate cryosurgery, or laser procedure;
* Neurological diseases or disorders affecting the bladder: Parkinson disease, multiple system atrophy, multiple sclerosis, spinal cord injury, cervical myelopathy, acute transverse myelitis, diabetic cystopathy, or dysfunctional voiding (non-neurogenic neurogenic bladder or Hinman syndrome);
* Psychiatric conditions: Participant has current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc.);
* Malignancy: Participant has a history of cancer (with the exception of skin cancer).

Control group exclusion criteria:

In addition to the exclusion criteria listed above, additional criteria for control subjects are as follows:

* Chronic Pain: In the past year, symptoms of discomfort or pain in the pelvic region for a period longer than 3 months within the preceding year;
* Infection: Volunteers who have had a urinary tract infection with a urine culture value of >100,000 colony forming units/ml (CFU/ml) within the past three months.
* Intravesical Therapy: Volunteers treated with intravesical chemotherapy or Bacillus Calmette-Guerin (BCG) therapy;
* Gastrointestinal Conditions: Volunteers with inflammatory bowel disease (such as Crohn's disease or ulcerative colitis, but not irritable bowel syndrome).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Microbiome | Within 6 month period from baseline evaluation
  Evaluate the microbiome at baseline, one "good day" (minimal or no symptoms) and one "bad day" (worst symptoms) within a 6 month period

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Burnett, MD, FACS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States